CLINICAL TRIAL: NCT05539235
Title: Efficacy and Safety of Intravitreal Conbercept With Modified Treat-and-Extend Regimens in Exudative Age-Related Macular Degeneration
Brief Title: Efficacy and Safety of Intravitreal Conbercept With Modified Treat-and-Extend Regimens in Exudative AMD
Acronym: IIT-A
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hui Peng, Chief Physician, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPeng
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Exudative age-related macular degeneration; anti-VEGF drug; Treat-and-extend; Conbercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Peng Hui, chief physician of Ophthalmology Department of the First Affiliated Hospital of Chongqing Medical University, randomly divided the enrolled patients into two groups when they only knew the patient number and did not know the specific situation of the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 week group (Experimental): Drug injection adjustment interval is 2 weeks
  Interventions: Drug: different degrees of adjustment of the injection interval
- 4 week group (Experimental): Drug injection adjustment interval is 4 weeks
  Interventions: Drug: different degrees of adjustment of the injection interval

INTERVENTIONS:
Drug: different degrees of adjustment of the injection interval — Treatment was an intravitreal injection of 0.5 mg conbercept using modified "T&E" treatment plans. After 3 months of monthly intravitreal injections, the patients were randomly divided into two groups, and the degree of adjustment of the injection interval was divided into 2 weeks and 4 weeks.
  Other Names: Modified Treat-and-Extend Regimens

SUMMARY:
This is a prospective study. Data from patients diagnosed with nAMD who have never received related treatment were collected. Treatment was an intravitreal injection of 0.5 mg conbercept using modified "T&E" treatment plans. After three months of monthly intravitreal injections, the patients were randomly divided into two groups, and the degree of adjustment of the injection interval was divided into two weeks and four weeks. Unlike the ALTAIR study, we cancel the maintenance criteria of classical T&E regimens. The best-corrected visual acuity (BCVA), central retinal thickness (CRT), last injection interval, and the number of injections were recorded at 3, 6, 12, and 24 months to evaluate treatment efficacy.

DETAILED DESCRIPTION:
This is a prospective study. Data from patients diagnosed with nAMD who have never received related treatment were collected. Treatment was an intravitreal injection of 0.5 mg conbercept using modified "T&E" treatment plans. After three months of monthly intravitreal injections, the patients were randomly divided into two groups, and the degree of adjustment of the injection interval was divided into two weeks and four weeks. Unlike the ALTAIR study, we cancel the maintenance criteria of classical T&E regimens. The best-corrected visual acuity (BCVA), central retinal thickness (CRT), last injection interval, and the number of injections were recorded at 3, 6, 12, and 24 months to evaluate treatment efficacy.

Randomization and Interventions Conbercept (0.5 mg) was injected intravitreally once a month for 3 months, and then the patients were randomly divided into a 2-week group and a 4-week group. 2-week group: The injection interval was adjusted to 2 weeks. 4-week group: The injection interval was adjusted to 4 weeks. In the 2-week group, if the visual acuity decreased by less than 5 letters and the lesions showed no signs of exudative activity, such as rebleeding and increased oedema, the patients were followed up 6 weeks after the third injection and injected intravitreally once. If the condition remained stable, the follow-up was extended to 8 weeks , vitreous infusion was performed, and then the vitreous injection interval was gradually extended. If visual acuity decreased by more than 5 letters or the lesions showed rebleeding, increased oedema and other anatomical indicators worsened, a 4-week injection interval was maintained or reduced to 2 weeks based on the extended injection interval. In the 4-week group, the patients were followed up 8 weeks after the third injection and injected intravitreally once. If the condition remained stable, the follow-up was extended to 12 weeks, and vitreous injection was performed. Then, the vitreous injection interval was gradually extended.

ELIGIBILITY:
Inclusion Criteria:

* age ≥50 years and meeting the diagnostic criteria for exudative AMD
* OCTA suggesting the presence of subretinal neovascularization
* no prior treatment (anti-VEGF, PDT, etc.)
* best-corrected visual acuity (BCVA) between 5-75 letters in the study eye.

Exclusion Criteria:

* allergy to drugs needed in the diagnosis and treatment
* a history of internal eye surgery (except surgery about cataract), trauma, or fundus laser photocoagulation
* other ophthalmologic diseases besides nAMD or cataracts
* renal insufficiency and severe cardiovascular and cerebrovascular diseases
* surgery required due to vitreous hemorrhage during follow-up treatment
* recent preparation for childbirth, pregnancy or lactation
* poor compliance with diagnosis and treatment or difficulty conducting a regular outpatient review and cooperating with treatment.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
mean change of the best-corrected visual acuity | baseline, every time before pre-intervention
  change of the best-corrected visual acuity

SECONDARY OUTCOMES:
mean change of central retinal thickness | baseline, every time before pre-intervention
  change of central retinal thickness
mean time of last injection interval | up to 2 years
  last injection interval
mean number of injections | up to 2 years
  number of injections
the rate of complications or adverse reactions | up to 2 years
  IOP, corneal epithelial defects, subconjunctival hemorrhage, secondary glaucoma, iatrogenic cataract, vitreous hemorrhage, endophthalmitis, systemic complications,

CONTACTS AND LOCATIONS:
Overall Officials: Hui Peng, PH.D, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
Results available in the paper after publication

REFERENCES:
- [Derived] Xie H, Ju H, Lu J, Wang X, Peng H. Comparative study on the efficacy of Conbercept and Aflibercept in the treatment of neovascular age-related macular degeneration. Sci Rep. 2024 May 25;14(1):11997. doi: 10.1038/s41598-024-62536-8. PMID 38796619